CLINICAL TRIAL: NCT06349889
Title: Adebrelimab Combined with Chemoradiotherapy for High-risk Locoregionally Advanced Nasopharyngeal Carcinoma: a Phase 2, Multicenter, Single-arm Clinical Trial
Brief Title: Adebrelimab and Chemoradiotherapy in High-risk LANPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NPC-II-004
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer
Keywords: immunotherapy; Chemoradiotherapy; PD-L1
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Adebrelimab 1200mg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 9 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — Drug: Adebrelimab Adebrelimab 1200mg will be given every 3 weeks for 3 cycles in induction chemotherapy and for 9 cycles in adjuvant chemotherapy, started on day 1 of induction chemotherapy and adjuvant chemotherapy, respectively.
  Other Names:
  PD-L1 antibody
  Drug: Gemcitabine Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
  Other Names:
  GEM
  Drug: Cisplatin Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
  Other Names:
  DDP
  Radiation: Intensity-modulated radiotherapy Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
  Other Names:
  IMRT

SUMMARY:
This trial aims to study the role of Adebrelimab combined with induction chemotherapy plus concurrent chemoradiotherapy (IC+CCRT) for high-risk locoregionally advanced nasopharyngeal carcinoma(LANPC).

DETAILED DESCRIPTION:
The trial plans to enroll patients with stage IVA+T3N2M0 (AJCC 8th) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Patients receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation plus Adebrelimab in induction chemotherapy and adjuvant chemotherapy. Adebrelimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 3 cycles in induction therapy and for 9 cycles in adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed nasopharyngeal carcinoma.
2. Tumor staged as IVA+T3N2M0 (AJCC 8th).
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug

Exclusion Criteria:

1. Age > 65 or < 18.
2. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
3. Hepatitis C virus (HCV) antibody positive
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
6. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
7. Has a known history of interstitial lung disease.
8. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
9. Is pregnant or breastfeeding.
10. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
11. Has known allergy to large molecule protein products or any compound of Adebrelimab.
12. Has a known history of human immunodeficiency virus (HIV) infection.
13. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  calculated from enrolment to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  calculated from enrolment to the date of death from any cause.
Distant metastasis-free survival (DMFS) | 3 years
  calculated from enrolment to the date of first distant metastasis.
Locoregional recurrence-free survival (LRRFS) | 3 years
  calculated from enrolment to the date of locoregional persistence or 1st locoregional recurrence.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | 3 years
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 13-16 weeks after radiotherapy, 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.
Failure-free survival (FFS) within different subgroups | 3 years
  analyses for FFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (≤4000copies/ml vs. >4000copies/ml), different Programmed Death-1（PD-L1） expression levels, age, gender, performance status, T category, N category, and stage (III vs. IVA).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.

REFERENCES:
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545